CLINICAL TRIAL: NCT00209092
Title: Randomized Phase II Trial of Sequential Docetaxel Followed by Capecitabine Versus Concomitant, Dose-Dense Docetaxel/Capecitabine as in Induction Therapy for Early Stage Breast Cancer
Brief Title: Randomized Phase II Trial Induction Therapy for Early Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Center for Oncology Research & Education (Other); Sanofi (Industry)
Responsible Party: Principal Investigator, Amelia Zelnak, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1114-2003
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential Therapy (Active Comparator): Docetaxel will be given at 100mg/m^2 intravenous Day 1 every 3 weeks for 4 cycles followed by capecitabine 1000 mg/m^2 twice a day by mouth Day 1-14 every 3 weeks for 4 cycles (total 8 cycles) (total 24 weeks).
  Interventions: Drug: Docetaxel; Drug: Capecitabine
- Concurrent Therapy (Active Comparator): Docetaxel will be given at 50mg/m^2 Intravenous Day1 concomitantly with capecitabine 1000 mg/m^2 twice a day by mouth Day 1-7 every 2 weeks for 8 cycles (total 16 weeks).
  Interventions: Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — Sequential Therapy: Docetaxel will be given at 100 mg/m^2 Intravenously (IV)Day 1 every 3 weeks for 4 cycles.
  Concurrent Therapy: Docetaxel will be given at 50 mg/m^2 IV Day 1.
Drug: Capecitabine — Sequential Therapy: administration of capecitabine 1000 mg/m^2 twice a day by mouth Day 1-14 every 3 weeks for 4 cycles (total 8 cycles) Concurrent Therapy: capecitabine 1000 mg/m^2 twice a day by mouth Day 1-7 every 2 weeks for 8 cycles (total 16 weeks).

SUMMARY:
The purpose of this study is to find out if the combination of docetaxel and capecitabine can shrink the size of breast tumors and preserve the breast.

DETAILED DESCRIPTION:
The purpose of this study is to identify new chemotherapy treatment regimens with better response rates and to find out if the combination of docetaxel and capecitabine can shrink the size of breast tumors and preserve the breast.

Induction chemotherapy offers the possibility of less surgery and determines tumor sensitivity in vivo. Previous trials have demonstrated that complete pathologic response in the breast at surgery corresponds with improved outcome. Additionally, we will correlate specific molecular markers in the breast tumors before and after chemotherapy, with response to treatment. Expression of these molecular markets may be used in the future to predict the likelihood of response to chemotherapy given post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast carcinoma.
* Early stage breast cancer (stage 1, 2, 3).
* No evidence of disease outside the breast or chest wall, except ipsilateral axillary lymph nodes.
* 18 years of age or older.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Prior chemotherapy, hormonal therapy, biologic therapy or radiation therapy for breast cancer.
* Major surgery within 28 days of study entry.
* Evidence of central nervous system (CNS) metastases.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Zelnak, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (19):
- United States (19):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Augusta Oncology Associates, PC 1348 Walton Way, Ste. 4300, Augusta, Georgia
  - Augusta Oncology Associates, PC 3696 Wheeler Road, Augusta, Georgia
  - WellStar Health System-Georgia Cancer Specialists, Austell, Georgia
  - WellStar Health System-Northwest Georgia Oncology Center, PC, Austell, Georgia
  - WellStar Health System-Northwest Georgia Oncology Center, PC, Carrollton, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Suburban Hematology-Oncology Associates, PC, Duluth, Georgia
  - South Atlanta Hematology-Oncology Group, East Point, Georgia
  - Suburban Hematology-Oncology Associates, PC, Lawrenceville, Georgia
  - Central Georgia Cancer Care, PC, Macon, Georgia
  - WellStar Health System-Georgia Cancer Specialists, Marietta, Georgia
  - WellStar Health System-Northwest Georgia Oncology Center, PC, Marietta, Georgia
  - South Atlanta Hematology-Oncology Group, Riverdale, Georgia
  - Suburban Hematology-Oncology Associates, PC, Snellville, Georgia
  - South Atlanta Hematology-Oncology Group, Stockbridge, Georgia
  - Central Georgia Cancer Care, PC, Warner Robins, Georgia

REFERENCES:
- [Result] Zelnak AB, Styblo TM, Rizzo M, Gabram SG, Wood WC, Harichand-Herdt S, Kim S, Liu Y, O'Regan RM; Georgia Center for Oncology Research and Education. Final results from phase II trial of neoadjuvant docetaxel and capecitabine given sequentially or concurrently for HER2-negative breast cancers. Clin Breast Cancer. 2013 Jun;13(3):173-9. doi: 10.1016/j.clbc.2012.12.004. Epub 2013 Jan 16. PMID 23332349
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A:Sequential Therapy: Docetaxel will be given at 100mg/m^2 intravenously Day1 every 3 weeks for 4 cycles followed by capecitabine 1000 mg/m^2 twice a day by mouth D1-14 every 3 weeks for 4 cycles (total 8 cycles) (total 24 weeks).
- Arm B:Concurrent Therapy: Docetaxel will be given at 50mg/m^2 intravenously Day 1 concomitantly with capecitabine 1000 mg/m^2 twice a day by mouth Day 1-7 every 2 weeks for 8 cycles (total 16 weeks).
Period: Overall Study
Arm/Group | Arm A:Sequential Therapy | Arm B:Concurrent Therapy
Started | 25 | 26
Completed | 17 | 24
Not Completed | 8 | 2
Not completed — Progression of disease | 7 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A:Sequential Therapy | Arm B:Concurrent Therapy | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 1 | 1
Age, Customized [Median (Full Range); unit: participants] | 50.8 [38 to 63] | 49.8 [29 to 66] | 50.3 [29 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Pathologic Response Rate to Pre-operative Treatment in Arm A (Docetaxel for 4 Cycles Followed by Capecitabine for 4 Cycles) or Arm B (Docetaxel + Capecitabine for 8 Cycles) in Patients With Early Stage Breast Cancer.
Description: Pathologic complete response (pCR): Absence of invasive breast cancer in the breast.
  Overall Clinical Response=Complete response(CR-complete disappearance of all measurable malignant disease)+partial response(PR-reduction by at least 30%)
  Stable disease (SD): No decrease or <25% increase in the sum of the products of the longest perpendicular diameters of all measurable lesions.
  Progressive disease (PD): A 20% or greater increase in a single lesion, OR reappearance of any lesion which has disappeared, OR clear worsening of any evaluable disease OR appearance of any new lesion/site.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Arm A:Sequential Therapy | Arm B:Concurrent Therapy
Number analyzed (Participants) | 25 | 26
participants
  Pathologic Complete Response-Overall population | 2 | 3
  Overall Clinical Response | 15 | 23
  Stable disease | 3 | 1
  Progressive Disease | 7 | 2

2. Secondary Outcome: Long Term Follow up Data on Recurrence and Survival
Description: Number of Patients remained alive and relapse free
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Arm A:Sequential Therapy | Arm B:Concurrent Therapy
Number analyzed (Participants) | 24 | 26
participants | 19 | 21

ADVERSE EVENTS:
Arm/Group | Arm A:Sequential Therapy | Arm B:Concurrent Therapy
Serious Adverse Events (participants affected / at risk) | 6/25 | 11/26
Other Adverse Events (participants affected / at risk) | 25/25 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A:Sequential Therapy (N=25) | Arm B:Concurrent Therapy (N=26)
Diarrhea (Gastrointestinal disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Neuropathy (Nervous system disorders) | 0 | 1
Hand and Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Liver Tests (Hepatobiliary disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Chest Pain (Cardiac disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A:Sequential Therapy (N=25) | Arm B:Concurrent Therapy (N=26)
Diarrhea (Gastrointestinal disorders) | 14 | 10
Neuropathy (Nervous system disorders) | 14 | 14
Neutropenia (Blood and lymphatic system disorders) | 2 | 8
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 14 | 18
Anemia (Blood and lymphatic system disorders) | 10 | 5
Fatigue (General disorders) | 20 | 17
Nausea (Gastrointestinal disorders) | 9 | 11
Anorexia (General disorders) | 5 | 5
Myalgias/Arthralgias (Musculoskeletal and connective tissue disorders) | 12 | 9
Hyperglycemia (Endocrine disorders) | 16 | 16
Liver Tests (Hepatobiliary disorders) | 10 | 9
Nail changes (Skin and subcutaneous tissue disorders) | 14 | 13
Muscositis (Gastrointestinal disorders) | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes